CLINICAL TRIAL: NCT05371080
Title: A Phase 3b, Open-label, Multi-country, Multi-centre, Long-term Follow-up Study of ZOSTER-049 (Follow-up of ZOSTER-006/022 Studies) to Assess the Prophylactic Efficacy, Safety and Persistence of Immune Response of a Herpes Zoster Subunit Vaccine and Assessment of Persistence of Immune Response and Safety of 1 or 2 Additional Doses Administered in ZOSTER-049 in 2 Subgroups of Older Adults
Brief Title: A Study on the Long-term Efficacy, Safety and Persistence of Immune Response of a Vaccine Against Herpes Zoster in Older Adults
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 217917; 2021-005319-30 (EudraCT Number)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Herpes Zoster
Keywords: Shingles; Herpes Zoster subunit vaccine; Recombinant Zoster Vaccine (RZV); Long-term follow-up study; Long-term vaccine efficacy; Prophylactic efficacy; Safety; Persistence of immune response; Older adults
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Intervention Model Description: Interventional study model and allocation in the current study follow the same approach as presented in the primary studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LTFU Group (Other): Participants who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and are followed for long-term vaccine efficacy and safety in the current ZOSTER-101 study.
  Interventions: Biological: HZ/su vaccine
- 1-Additional Dose Group (Other): Participants who received two doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies and one additional dose of the HZ/su vaccine in the ZOSTER-049 study and are followed for persistence of immunogenicity and safety in the current ZOSTER-101 study.
  Interventions: Biological: HZ/su vaccine
- Revaccination Group (Other): Participants who received two doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies and two additional doses of the HZ/su vaccine in the ZOSTER-049 study and are followed for persistence of immunogenicity and safety in the current ZOSTER-101 study.
  Interventions: Biological: HZ/su vaccine
- Control Group (Other): Participants who received two doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the ZOSTER-049 study, but who served as a control for the two groups that received 1 or 2 additional doses of HZ/su (1-Additional Dose and Revaccination groups). In the current ZOSTER-101 study, this Control group is used in the evaluation of the long-term vaccine efficacy, safety and as a control for persistence of immunogenicity to additional doses administered in ZOSTER-049 study.
  Interventions: Biological: HZ/su vaccine

INTERVENTIONS:
Biological: HZ/su vaccine — No study intervention is administered in this extension study. Participants received the HZ/su vaccine administered in the ZOSTER-049 (NCT02723773), ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) primary studies. In order to assess the persistence of immune responses, participants provide blood samples at Day 1 and yearly from Month 12 until Month 48 in the current ZOSTER-101 study, according to their study group assignment. In case of a suspected HZ case diagnosis in any of the participants, clinical specimens from HZ lesions (3 replicate samples, collected on the same day, per participant) are collected to confirm the diagnosis of HZ by Polymerase Chain Reaction (PCR)

SUMMARY:
The purpose of the current ZOSTER-101 long-term follow-up (LTFU) study of ZOSTER-049 (NCT02723773) study, an extension of ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) primary studies, is to assess the long-term vaccine efficacy (VE) against Herpes Zoster (HZ) (approximately 11-15 years post primary vaccination in ZOSTER-006/022 studies), persistence of immunogenicity and safety of GSK's Herpes Zoster subunit (HZ/su) vaccine in older adults. The persistence of immunogenicity and safety of 1 or 2 additional doses (0, 2-month schedule) of HZ/su vaccine administered to a small group of participants in ZOSTER-049 study (approximately 5 years after the initial vaccination in ZOSTER-006/022 studies) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants and participant's caregiver, who, in the opinion of the investigator, can and are willing to comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Medically stable participants as established by medical history and clinical examination before entering into the study.
* Participants who completed ZOSTER-049 study (following at least 1 dose of HZ/su in ZOSTER-006/022 studies).

Exclusion Criteria:

Medical conditions

* Any clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) for the treatment of HZ or Varicella Zoster Virus (VZV) infection at the time of enrolment or their planned use during the study period.
* Previous vaccination against VZV or HZ and/or planned administration during the study of a VZV or HZ vaccine (including an investigational or non-registered vaccine other than HZ/su administered in studies ZOSTER-006/022 or ZOSTER-049).

Prior/Concurrent clinical study experience

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device) for the prevention and/or treatment of HZ or VZV and which may have a possible activity against VZV.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3038 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2027-08-23 (Estimated); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
Number of participants in LTFU and Control groups with confirmed HZ cases | During the total duration of ZOSTER-101 study (Day 1 through Month 48)
  A suspected case of HZ is defined as new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) and no alternative diagnosis.
  A suspected case of HZ can be confirmed in two ways:
  * By PCR;
  * By the HZ Ascertainment Committee (HZAC).

SECONDARY OUTCOMES:
Number of participants in LTFU and Control groups with confirmed HZ cases | From 1-month post-Dose 2 in the ZOSTER-006/022 studies until the end of the ZOSTER-101 study at Month 48
  A suspected case of HZ is defined as new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) and no alternative diagnosis.
  A suspected case of HZ can be confirmed in two ways:
  * By PCR;
  * By the HZAC.
Anti-glycoprotein E (gE) antibody concentrations | At Day 1, Months 12, 24, 36 and 48 in the ZOSTER-101 study
  Anti-gE antibody concentrations are expressed as geometric mean concentrations (GMCs), as determined by enzyme-linked immunosorbent assay (ELISA).
Frequency of gE-specific Cluster of Differentiation (CD)4+ T-cells secreting at least two activation markers from among IFN-γ, IL-2, TNF-α, CD40L | At Day 1, Months 12, 24, 36 and 48 in the ZOSTER-101 study
Percentage of participants with serious adverse events (SAEs) causally related to the study intervention | During the total duration of the ZOSTER-101 study (Day 1 through Month 48)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, or results in disability/incapacity. Relationship between study intervention and the occurrence of SAEs is assessed by the investigator using clinical judgement.
Percentage of participants with potential immune-mediated diseases (pIMDs) (serious and non-serious) causally related to the study intervention | During the total duration of the ZOSTER-101 study (Day 1 through Month 48)
  pIMDs are a subset of adverse events of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. A serious pIMD is any pIMD that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, or results in disability/incapacity. Relationship between study intervention and the occurrence of pIMDs is assessed by the investigator using clinical judgement.
Percentage of participants with HZ-related complications of confirmed HZ | During the total duration of the ZOSTER-101 study (Day 1 through Month 48)
  A suspected case of HZ is defined as new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) and no alternative diagnosis.
  A suspected case of HZ can be confirmed in two ways:
  * By PCR;
  * By the HZAC. HZ complications are the following: post-herpetic neuralgia, HZ vasculitis, disseminated disease, ophthalmic disease, neurologic disease, visceral disease or stroke A.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (95):
- United States (8):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Australia (3):
  - GSK Investigational Site, Warrawong, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Geelong, Victoria
- Brazil (3):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, São Paulo
- Canada (8):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Hradec Králové
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (5):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Rosiers-d'Égletons
- Germany (15):
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Shatin, Hong Kong
- Italy (2):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Durango, Mexico
- South Korea (5):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Balenyà (Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, La Roca del Vallès
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda( Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Peralada( Girona)
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic
- Sweden (9):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Upplands Vasby
  - GSK Investigational Site, Uppsala
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan
- United Kingdom (5):
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Bradford-on-Avon, Wiltshire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Broughshane
  - GSK Investigational Site, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.